CLINICAL TRIAL: NCT07306611
Title: Regenerative Treatment of Female Genital Atrophy
Acronym: RETREAT-FUGA
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: AndreiaAntunes (Other)
Collaborators: Portuguese National Funding Agency for Science, Research and Technology (FCT) (Unknown); University of Minho (Other); Hospital Santo André - Centro Hospitalar de Leiria (Unknown)
Responsible Party: Sponsor-Investigator, AndreiaAntunes, affiliated investigator, PhD Student, Consultant of Gynecology and Obstetrics, Instituto Politécnico de Leiria
Organization: Instituto Politécnico de Leiria (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 27/2024 CE ULS-RL; PHD SCHOLARSHIP 2021. 07973.BD (Other Grant/Funding Number: Portuguese Foundation for Science and Technology)
Record Dates: First submitted 2025-12-14; First posted 2025-12-29 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Vulvo Vaginal Atrophy
Keywords: Vulvovaginal atrophy; menopause; Ageing; regenerative treatment; platelets-rich plasma; autologous plasma
MeSH Terms: interventions — Mesotherapy; Saline Solution

STUDY DESIGN:
Intervention Model Description: The sample is adult women aged 25-80 years followed at the gynecology appointment of ULS RL.
  Potential participants (n= 30) were enrolled at specific gynecology consultation of genital atrophy at the ULS RL. We considered an N=30 because this is the minimum number of individuals according to the central limit theorem to obtain a normal Gaussian distribution of the sample.
  This was a randomized controlled trial using a random number table in two treatment groups (PRP versus placebo-saline solution), Participants were randomized in a 3:2 ratio to receive either the active treatment or placebo. A computer-generated randomization list containing 30 assignments (18 treatment and 12 placebo) was created using simple randomization without replacement. Each participant was assigned the next sequence was generated before participant enrollment and kept concealed from investigators.
  Several measures were collected to obtaining statistically robust estimates.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PRP Group (Active Comparator): GROUP A (18 patients) random assign from enrolled patients: Participants receive intradermal injections of autologous platelet-rich plasma (PRP) into the vulvar vestibule, followed by topical application of platelet-poor plasma (PPP) gel for 5 days.
  Interventions: Biological: Mesotherapy with Autologous Platelet-Rich Plasma (PRP) to vulvovaginal area; Biological: Platelet-Poor Plasma Gel
- Placebo Group (Placebo Comparator): GROUP B (12 patients) random assign from enrolled patients: Participants receive intradermal injections of saline solution into the vulvar vestibule, followed by topical application of platelet-poor plasma (PPP) gel for 5 days.
  Interventions: Other: Mesotherapy with saline solution; Biological: Platelet-Poor Plasma Gel

INTERVENTIONS:
Biological: Mesotherapy with Autologous Platelet-Rich Plasma (PRP) to vulvovaginal area — Intervention: Autologous Platelet-Rich Plasma Injection Type: Biological Description: Autologous PRP is prepared from peripheral venous blood collected into sterile citrate-containing PRP tubes with cell-separator gel. Samples are centrifuged at 3400 rpm (1200 g) for 7 minutes at room temperature. Platelet-poor plasma (PPP) is separated and activated with calcium gluconate to obtain a topical gel. PRP is obtained by releasing platelets from the gel and aspirating the platelet-enriched plasma. After vulvar disinfection and topical anesthesia, 2 ml of PRP is injected intradermally using a 27-gauge, 13 mm needle. Six injections are administered along the vulvar vestibule (anterior, posterior, and bilateral lateral sites) using a linear retrograde technique. Local compression is applied for one minute. Participants apply PPP gel twice daily for 5 days.
  Arms: PRP Group
Other: Mesotherapy with saline solution — Description: Participants receive intradermal injections of 2 ml sterile saline solution into the vulvar vestibule following the same injection sites, technique, needle size, and procedural steps as the PRP group. Six injections are administered using a linear retrograde technique, followed by local compression and topical PPP gel application twice daily for 5 days.
  Arms: Placebo Group
Biological: Platelet-Poor Plasma Gel — Description: Activated platelet-poor plasma gel is applied topically to the vulvar area using a cotton swab twice daily for five days following the procedure. This intervention is administered to participants in both study arms

SUMMARY:
Vulvovaginal health is a key aspect of active and healthy aging for all women. Hormonal deprivation that occurs during menopause significantly affects the anatomy and function of urogenital tissues, leading to their atrophy. Vaginal creams and suppositories containing estrogens are the standard treatment and can improve this condition. However, they require continuous application, which often makes adherence to treatment challenging. Additionally, women with hormone-dependent tumors, such as most breast cancers and many gynecological cancers, are even more affected by this issue. These women are often treated with anti-estrogen medications, undergo radio or chemotherapy, and are frequently younger, with the added complication that the standard treatment is contraindicated for them.

To address this important issue, the study titled "Regenerative Treatment of Female Genital Atrophy" was developed. If you meet the required criteria, we would like to invite you to participate.

Inclusion Criteria:

* Clinical complaints of genital atrophy (e.g., dryness, burning, itching, discomfort, or pain during intercourse).
* Contraindication to standard local hormonal treatment (e.g., allergy, bothersome side effects, lack of improvement with standard treatment, history of hormone-dependent cancer, or thrombotic event treated at least two years ago).

This study focuses on Regenerative Medicine, which aims to support the regeneration of cells, tissues, or organs in the human body to restore normal function. This field holds significant curative and preventive potential. The selected regenerative treatment, widely used in various medical fields (such as dentistry and orthopedics), is derived from the patient's own body, making it a natural and safe option with minimal side effects. This treatment, known as platelet-rich plasma (PRP), has shown effectiveness in improving the firmness, elasticity, hydration, and thickness of the vulva and vagina. However, further research is required to assess the effectiveness of PRP specifically in the external female genital area.

What is PRP - Platelet-Rich Plasma? PRP is a substance obtained from the patient's own blood. Blood is composed of several components, including red blood cells, white blood cells, plasma, and platelets. Platelets are small cell fragments that play a crucial role in blood clotting and wound healing. PRP is created by taking a small sample of the patient's blood and processing it in a centrifuge to concentrate the platelets within the plasma. This concentrated plasma, rich in growth factors and proteins, is then injected into the target area to stimulate tissue regeneration and repair. Because PRP is derived from the patient's own body, it is considered a natural and safe treatment with a very low risk of adverse reactions.

PRP is obtained by collecting a small amount of the patient's blood. After a carefully standardized preparation process, the PRP is injected into the vulvovaginal area under local anesthesia.

Study Location: Gynecology Department of Santo André Hospital, Leiria, at the Genital Atrophy Clinic.

Study Protocol:

* Initial evaluation consultation.
* First treatment intervention.
* Follow up approximately one month after the first treatment and second treatment intervention.
* Another follow-up approximately one month after the second treatment.
* Final evaluation six months after the start of the study. Participants are divided into two groups: one group receives PRP treatment, while the other receives a placebo (serum). At the end of the study, participants in the placebo group will have the option to undergo PRP treatment.

This is a double-blind study designed to evaluate the efficacy of PRP in the female external genital area.

DETAILED DESCRIPTION:
Introduction:

Vulvovaginal atrophy (VVA) is a condition associated with lower urinary tract dysfunction caused by decreased levels of estrogen and androgens, collectively referred to as genitourinary syndrome of menopause (GSM). Approximately 50% of postmenopausal women experience symptoms related to urogenital atrophy, which significantly impacts sexual function and quality of life (QoL) worldwide. These symptoms include vaginal dryness, irritation, dyspareunia, and recurrent infections, leading to discomfort, reduced intimacy, and emotional distress.

VVA symptoms are associated with decrements in quality of life that may be comparable to serious conditions such as arthritis, chronic obstructive pulmonary disease, asthma, and irritable bowel syndrome.

Contrary to vasomotor symptoms of menopause, which tend to diminish over time, GSM symptoms often worsen, leading to a greater impact on QoL and negatively affecting patients' confidence and intimacy with their partners. Current standard treatments, such as low-dose vaginal estrogens, are effective in alleviating symptoms but require continuous application, which can hinder adherence. Furthermore, these treatments are contraindicated in women with hormone-dependent cancers or a history of thrombotic events, leaving a significant population without effective therapeutic options.

Regenerative options include injection of materials into the vaginal such as PRP, fat graft, hyaluronic acid, botulinum toxin, and collagen, seems promising options, but to date their efficacy has not been reviewed, so further studies are required, and the procedures should be standardized to benefit more patients.

PRP is the most common autologous regenerative treatment used in different medical fields (maxillo-facial, dermatology, cardiac surgery, pediatric surgery, gynecology, urology, plastic surgery, and ophthalmology)and poses a low risk adverse events.

Platelets contain an abundance of growth factors and cytokines that can affect inflammation, angiogenesis, stem cell migration, and cell proliferation. Based on histological evidence, PRP injected in human deep dermis and sub-cutaneous tissue induces soft-tissue augmentation, activation of fibroblasts, and new collagen deposition, as well as new blood vessels and adipose tissue formation, induction of dermal collagenases, angiogenesis, and adipogenesis in human skin by injection of platelet-rich fibrin matrix. PRP is more than just a platelet concentrate; it also contains proteins to cell adhesion that allow the use of PRP product into a biologic gel cream for surface application.

Objectives:

The primary objective of this study is to evaluate the efficacy and safety of autologous PRP for the treatment of VVA in women with contraindications or inefficacy to local hormonal treatments. Specifically, the study aims to:

1. Assess the ability of PRP to restore vaginal tissue integrity, including firmness, elasticity, hydration, and thickness.
2. Evaluate the improvement of VVA symptoms, such as dryness, irritation, and dyspareunia.
3. Measure the impact of PRP treatment on patients' quality of life and sexual function.
4. Monitor and document any adverse effects associated with PRP treatment.

Study Protocol:

Participants will be randomly assigned to one group:

1. PRP Group: Patients will receive autologous PRP injections into the vulvovaginal area.
2. Placebo Group: Patients will receive placebo (saline solution) injections.

The study will follow a standardized protocol:

* T0 (Baseline): Initial evaluation, including medical history, gynecological examination, and baseline symptom assessment.
* T1 (1 Month): First treatment session.
* T2 (2 Months): Follow-up and second treatment session.
* T3 (3 Months): Follow-up evaluation.
* T4 (6 Months): Final evaluation, including symptom assessment, quality of life questionnaires, and laboratory tests.

Data Collection

Data will be collected at multiple times (T0, T1, T2, T3, and T4) using both clinical assessments and patient-reported outcome measures (PROMs). The following variables and tools will be used:

1. - Clinical Report Form (CRF):

   * Demographic and Health Data: Age, years since menopause, education level, occupation, body mass index (BMI), smoking habits, parity, medical history, current medications, and history of hormonal treatments.
   * Gynecological Examination:

   Visual assessment of the perineum, vulva, and vagina for signs of atrophy (e.g., pallor, petechiae, friability, narrowing of the vaginal opening).

   Cotton swab test to assess tissue sensitivity. Vaginal opening flexibility, measured in centimeters. Vulvovaginal Visual Examination Tool (VVET): A validated scale to assess vulvovaginal health, including color, epithelial integrity, surface thickness, and secretions. These ratings were summed and re-scaled to range from 0 to 12 to create a vaginal exam composite index. A score of 0 indicates normal vulva-vaginal characteristics and higher scores indicate greater degrees of vulva-vaginal atrophy
2. - Laboratory Investigations:

   * Vaginal Maturation Index (VMI): Cytological analysis of epithelial cells to assess atrophy.
   * Vaginal Maturation Value (VMV): Calculated using the formula: (0.2 × % parabasal cells) + (0.6 × % intermediate cells) + (1.0 × % superficial cells). A VMV ≤50 indicates atrophy.
   * Vaginal pH: Measured using pH strips, with values <5 indicating normal hormonal patterns.
3. - Patient-Reported Outcome Measures (PROMs):

   * Patient self-assessed symptoms of vulva and vaginal atrophy (VVA)• Vaginal • Vaginal and/or vulva irritation/itching/discomfort (none, mild, moderate or severe) • Dysuria/pain with urination (none, mild, moderate or severe) • Vaginal pain associated with sexual activity/pain with sex (none, mild, moderate or severe) • Vaginal bleeding associated with sexual activity (presence vs. absence) and identification of the most bothersome symptom.
   * EQ-5D: A generic instrument for measuring health-related quality of life, validated for European Portuguese.
   * Female Sexual Function Index (FSFI-6): A validated questionnaire assessing six domains of sexual function: desire, arousal, lubrication, orgasm, satisfaction, and pain.
   * The King´s Health Questionnaire (KHQ) assesses the impact of urinary incontinence on the QoL.
   * Day-to-Day Impact of Vaginal Aging (DIVA): A self-report measure of the impact of vaginal symptoms on daily life, emotional well-being, and sexual function.
   * Visual Analog Scale (VAS): Used to assess pain and discomfort during and after treatment.
   * Side Effects Questionnaire: Participants will report any side effects (e.g., pain, swelling, bruising) one week after each treatment.
   * Satisfaction Questionnaire: At the final visit (T4), participants will rate their overall satisfaction with the treatment and perceived improvement compared to baseline.

Feasibility: After each treatment, the co-investigator will be asked to evaluate the ease of treatment using a 5-point Likert scale.

Safety Measures

The safety of PRP treatment will be closely monitored throughout the study. Participants will be asked to document any side effects in a daily diary and report them during follow-up visits or phone interviews. The most common expected side effects include:

* Localized pain or discomfort.
* Swelling or edema.
* Bruising at the injection site. These side effects are expected to be mild, temporary, and self-limiting. Serious adverse events are not anticipated based on previous studies of PRP in gynecological and other medical applications.

Adverse Events Monitoring All adverse events will be documented in the source documents and the patient report form (PRF). The clinical course of each event will be followed until resolution or stabilization. If a participant experiences significant discomfort during the procedure (measured using the Visual Analog Scale), the intervention will be suspended, and appropriate medical care will be provided.

Participants will have access to the principal investigator via phone or email for immediate reporting of any concerns or adverse events.

Goals:

Primary endpoints Goal 1: The efficacy analyses demonstrate a statistically significant improvement from baseline T0 to T4, of treatment in following parameters: 1. Maturation Index of vaginal cytology (decrease of parabasal vulvovaginal cells and increase in superficial cells) 2. Lowering of the vaginal PH.

Goal 2: A statistically significant improvement of VVA symptoms self-identified by subjects as the most bothersome VVA symptom to her at baseline.

Goal 3: A statistically significant improvement of quantitative assessment of genital health with the VVET scale.

Secondary endpoints Secondary efficacy variables include the significant improvement of the other symptoms of VVA self-assessed by questionnaires and satisfaction with the treatment evaluated by the significant improve in the quality of life evaluated with several dimensional PROMs.

Ethical Considerations This study will be conducted in accordance with the Declaration of Helsinki, Good Clinical Practice (GCP) guidelines, and relevant European and Portuguese legislation. Ethical approval will be obtained from the Ethics Committee of Santo André Hospital and the Ethics Subcommittee for Life and Health Sciences of the University of Minho.

Informed Consent All participants will provide written informed consent before enrollment. They will be informed about the study objectives, procedures, potential risks, and benefits. Participants will have the right to withdraw from the study at any time without any impact on their medical care.

Confidentiality Participant confidentiality will be strictly maintained. Personal data will be anonymized and stored securely in password-protected systems and locked cabinets. Only authorized personnel will have access to identifiable information. Data will be managed in compliance with the EU General Data Protection Regulation (GDPR) and Portuguese Law nº 58/2019.

Harms The suspension of the intervention will occur through the verification of significant levels of discomfort during the procedure (Visual Analogue Scale). In case of events occurrence such as urinary tract infection, vulvovaginitis, irritation and vaginal injury after treatment. In these cases, an appropriate medical treatment will be offered. Nevertheless, we don´t expect any serious harms according to previous studies, being the most expected; pain, swelling or hematoma all of it temporary and auto limited.

Minorities This study intends to include all eligible women regardless of race, ethnic origin, or sexual orientation. VVA has been well studied in the USA, Europe, the Mid East, and Asian countries. A review of the literature has not revealed any differences in either diagnosis or treatment effects between racial or ethnic groups. The study is a preliminary investigation of regenerative treatment effects of PRP graft in all women pooled, regardless of ethnic or racial group.

Financial Issues and Resources

This study will not impose additional costs on the participating institution or patients. The following resources will be provided free of charge:

* Consumables (e.g., anesthetics, syringes, blood collection tubes, pH strips).
* Laboratory services for cytology and platelet count analysis. The estimated cost of the study is €6,000, which will be covered by the research team through funding from the Portuguese Science and Technology Foundation - FCT Medical PhD Scholarship and other sources.

Conflict of Interest The researchers declare no conflicts of interest related to the implementation of this study.

Communication and Use of Results

The results of this study will be disseminated through:

* Presentations at national and international scientific conferences.
* Publications in peer-reviewed scientific journals.
* Inclusion in the principal investigator's doctoral thesis. If the study yields positive results, it may serve as a basis for a Phase 3 clinical trial, contributing to the development of new therapeutic options for VVA with minimal environmental impact.

ELIGIBILITY:
Inclusion Criteria:

* At least one clinical complaint of VVA.

  * Dryness
  * Burning
  * Itching
  * Discomfort (soreness, irritation)
  * Dyspareunia (sexual impaired function)
  * With or without urinary problems (incontinence, urgency, dysuria). Must report a contra-indication with the standard local hormonal treatment.
  * Allergy
  * Burden side effects
  * Non-improvement with standard treatment
  * Hormonal cancer survivors must be in remission for two years after the last oncologic treatment.
  * Thrombotic disease patients must have the disease controlled and have passed 2 years after the thrombotic event.

Must have a cervicovaginal cytology confirming the atrophy, having ≤ 5% of superficial cells on vaginal smear. Moreover, a normal morphologic cytology besides the inflammatory or atrophy change is mandatory.

Must have a vaginal pH above 5 at baseline. Must have a normal mammography (American College of Radiology BI-RADS 1 or 2) within 12 months of study starts (Day 1), and normal breast examination.

Willing to participate in the study and sign an informed consent.

Exclusion Criteria:

* Life expectancy < 6 months due to concomitant illnesses.
* Exposure to any investigational drug or procedure within 1 month prior to study entry or enrolled in a concurrent study that may confound results of this study.
* Active infectious disease. Patients known to have tested positive for HIV, HTLV, HBV, HCV, CMV (IgM > IgG) and/or syphilis will have an expert consultation as to patient eligibility based on the patient's infectious status.
* Any illness which, in the Investigator's judgment, will interfere with the patient's ability to comply with the protocol, compromise patient safety, or interfere with the interpretation of the study results.
* Patients on chronic immunosuppressive transplant therapy.
* Known drug or alcohol dependence or any other factors which will interfere with the study conduct or interpretation of the results or who in the opinion of the investigator are not suitable to participate.
* Used oral, transdermal, vaginal, intrauterine, implants/injectables drugs that contained either oestrogens, progestins, androgens, or selective oestrogen receptor modulators (SERMs) before the study (a washout period of 4 weeks is required). Use of prescription and non-prescription medications and remedies known to alleviate VVA, discomfort including vaginal lubricants and moisturizers, are allowed during the study.
* Any allergic reaction to local anaesthetics.
* Unwilling and/or not able to give written informed consent.

Ages: 25 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2024-06-04 (Actual); Primary Completion 2025-06-18 (Actual); Study Completion 2025-11-26 (Actual)

PRIMARY OUTCOMES:
Efficacy of PRP treatment | • T0 (Baseline): Initial evaluation • T1 (1 Month): 1ª treatment. • T2 (2 Months): 2º treatment. • T3 (3 Months): Follow-up evaluation • T4 (6 Months): Final evaluation, including symptom assessment, quality of life questionnaires, and laboratory tests.
  Using SPSS software (version 26.0), the following statistical methods will be applied:
  * Descriptive Statistics: Means, standard deviations, frequencies, and percentages will summarize demographic and clinical characteristics.
  * Linear Mixed Models (LMMs): Used to evaluate changes in outcomes over time, controlling for assessment time and baseline characteristics. Adjusted means and 95% confidence interval.
  * Significance Testing: A p-value <0.05 will be considered statistically significant.
  * Effect Size: Standardized treatment effect will be calculated as the mean difference in change between T0 and T4, divided by the standard deviation (SD) of that difference. Effect sizes will be categorized as small (0.2), medium (0.5), or large (0.8).
  A statistically significant improvement of VVA symptoms self-identified by subjects at baseline and a significant perception of improvement of quantitative assessment of genital health with the VVET scale .

SECONDARY OUTCOMES:
Validation of a clinical Tool to visually classifying the severity of VVA and the characterization of the vulvovaginal area. | • T0 (Baseline): Initial evaluation • T3 (3 Months): Follow-up evaluation. • T4 (6 Months): Final evaluation
  A validated scale to assess vulvovaginal health, including color, epithelial integrity, surface thickness, and secretions.The original 4-point scale (0-none, 1-mild, 2-moderate, and 3-severe) was tested and adapted by the authors to an easier classification in three parameters (0-normal, 1-moderate change, 2-severe change) to assess parameters of vulvovaginal color, vaginal epithelial integrity, vaginal epithelial surface thickness, and vaginal secretions. These ratings were summed and rescaled to range from 0 to 12 to create a vaginal exam composite index. A score of 0 indicates normal vulvovaginal characteristics and higher scores indicate greater degrees of vulvovaginal atrophy. This task will intent to contribute for the validation of the selected visual scale to be use in research to reduce development costs, ease regulatory approval, and as a practical tool in clinical settings.

CONTACTS AND LOCATIONS:
Overall Officials: Andreia R Antunes, PhD Student and Medical Doctor, Principal Investigator — Minho University Medical School, ICVS - Life and Health Sciences Research Institute, IPL - Polytechnic University of Leiria, CitechCare - Center for Innovative Care and Health Technology, Local Health Unit of Leiria Region, Santo André Hospital; Maria S Guarino, PhD, Study Director — IPL - Polytechnic University of Leiria, CitechCare - Center for Innovative Care and Health Technology; Cristina Isabel Nogueira-Silva, PhD, Medical Doctor, Study Director — Minho University Medical School, ICVS - Life and Health Sciences Research Institute
Locations (1):
- Santo André Hospital, Leiria, Leiria District, Portugal

IPD SHARING:
Plan to Share IPD: No
Participants data will not be shared because study includes sensitive clinical information with a high risk of re-identification and current institutional and regulatory constraints do not permit external data sharing.

REFERENCES:
- [Background] Pinkerton JV, Shifren JL, La Valleur J, Rosen A, Roesinger M, Siddhanti S. Influence of raloxifene on the efficacy of an estradiol-releasing ring for treating vaginal atrophy in postmenopausal women. Menopause. 2003 Jan-Feb;10(1):45-52. doi: 10.1097/00042192-200310010-00008. PMID 12544676
- [Background] Greendale GA, Zibecchi L, Petersen L, Ouslander JG, Kahn B, Ganz PA. Development and validation of a physical examination scale to assess vaginal atrophy and inflammation. Climacteric. 1999 Sep;2(3):197-204. doi: 10.3109/13697139909038062. PMID 11910597
- [Background] Raymundo N, Yu-cheng B, Zi-yan H, Lai CH, Leung K, Subramaniam R, Bin-rong C, Ling YS, Nasri N, Calimon N. Treatment of atrophic vaginitis with topical conjugated equine estrogens in postmenopausal Asian women. Climacteric. 2004 Sep;7(3):312-8. doi: 10.1080/13697130400003147. PMID 15669556
- [Background] McCormack HM, Horne DJ, Sheather S. Clinical applications of visual analogue scales: a critical review. Psychol Med. 1988 Nov;18(4):1007-19. doi: 10.1017/s0033291700009934. PMID 3078045
- [Background] Huang AJ, Gregorich SE, Kuppermann M, Nakagawa S, Van Den Eeden SK, Brown JS, Richter HE, Walter LC, Thom D, Stewart AL. Day-to-Day Impact of Vaginal Aging questionnaire: a multidimensional measure of the impact of vaginal symptoms on functioning and well-being in postmenopausal women. Menopause. 2015 Feb;22(2):144-54. doi: 10.1097/GME.0000000000000281. PMID 24983271
- [Background] Viana R, Viana S, Neto F, Mascarenhas T. Adaptation and validation of the King's Health Questionnaire in Portuguese women with urinary incontinence. Int Urogynecol J. 2015 Jul;26(7):1027-33. doi: 10.1007/s00192-015-2628-6. Epub 2015 Feb 5. PMID 25653033
- [Background] Ferreira PL, Ferreira LN, Pereira LN. [Contribution for the validation of the Portuguese version of EQ-5D]. Acta Med Port. 2013 Nov-Dec;26(6):664-75. Epub 2013 Dec 20. Portuguese. PMID 24388252
- [Background] Ettinger B, Hait H, Reape KZ, Shu H. Measuring symptom relief in studies of vaginal and vulvar atrophy: the most bothersome symptom approach. Menopause. 2008 Sep-Oct;15(5):885-9. doi: 10.1097/gme.0b013e318182f84b. PMID 18779677
- [Background] Weber MA, Limpens J, Roovers JP. Assessment of vaginal atrophy: a review. Int Urogynecol J. 2015 Jan;26(1):15-28. doi: 10.1007/s00192-014-2464-0. Epub 2014 Jul 22. PMID 25047897
- [Background] Simon JA, Archer DF, Kagan R, Bernick B, Graham S, Constantine GD, Mirkin S. Visual improvements in vaginal mucosa correlate with symptoms of VVA: data from a double-blind, placebo-controlled trial. Menopause. 2017 Sep;24(9):1003-1010. doi: 10.1097/GME.0000000000000880. PMID 28419068
- [Background] Harrison P; Subcommittee on Platelet Physiology. The use of platelets in regenerative medicine and proposal for a new classification system: guidance from the SSC of the ISTH. J Thromb Haemost. 2018 Sep;16(9):1895-1900. doi: 10.1111/jth.14223. Epub 2018 Aug 11. PMID 30099839
- [Background] Turner L. ISSCR's Guidelines for Stem Cell Research and Clinical Translation: Supporting development of safe and efficacious stem cell-based interventions. Stem Cell Reports. 2021 Jun 8;16(6):1394-1397. doi: 10.1016/j.stemcr.2021.05.011. Epub 2021 May 27. PMID 34048693
- [Background] Hovatta O, Stojkovic M, Nogueira M, Varela-Nieto I. European scientific, ethical, and legal issues on human stem cell research and regenerative medicine. Stem Cells. 2010 Jun;28(6):1005-7. doi: 10.1002/stem.436. No abstract available. PMID 20533567
- [Background] Dawood AS, Salem HA. Current clinical applications of platelet-rich plasma in various gynecological disorders: An appraisal of theory and practice. Clin Exp Reprod Med. 2018 Jun;45(2):67-74. doi: 10.5653/cerm.2018.45.2.67. Epub 2018 Jun 29. PMID 29984206
- [Background] Varghese J, Acharya N. Platelet-Rich Plasma: A Promising Regenerative Therapy in Gynecological Disorders. Cureus. 2022 Sep 10;14(9):e28998. doi: 10.7759/cureus.28998. eCollection 2022 Sep. PMID 36249659
- [Background] Streit-Cieckiewicz D, Kolodynska A, Futyma-Gabka K, Grzybowska ME, Golacki J, Futyma K. Platelet Rich Plasma in Gynecology-Discovering Undiscovered-Review. Int J Environ Res Public Health. 2022 Apr 26;19(9):5284. doi: 10.3390/ijerph19095284. PMID 35564681
- [Background] Tsepkolenko A, Tsepkolenko V, Dash S, Mishra A, Bader A, Melerzanov A, Giri S. The regenerative potential of skin and the immune system. Clin Cosmet Investig Dermatol. 2019 Jul 15;12:519-532. doi: 10.2147/CCID.S196364. eCollection 2019. PMID 31410045
- [Background] White C, Brahs A, Dorton D, Witfill K. Platelet-Rich Plasma: A Comprehensive Review of Emerging Applications in Medical and Aesthetic Dermatology. J Clin Aesthet Dermatol. 2021 Nov;14(11):44-57. PMID 34980960
- [Background] Goldstein AT, Mitchell L, Govind V, Heller D. A randomized double-blind placebo-controlled trial of autologous platelet-rich plasma intradermal injections for the treatment of vulvar lichen sclerosus. J Am Acad Dermatol. 2019 Jun;80(6):1788-1789. doi: 10.1016/j.jaad.2018.12.060. Epub 2019 Jan 11. No abstract available. PMID 30639885
- [Background] Yano K, Watanabe N, Tsuyuki K, Ikawa T, Kasanuki H, Yamato M. Regulatory approval for autologous human cells and tissue products in the United States, the European Union, and Japan. Regen Ther. 2014 Nov 11;1:45-56. doi: 10.1016/j.reth.2014.10.001. eCollection 2015 Jun. PMID 31589662
- [Background] Coulange Zavarro A, De Girolamo L, Laver L, Sanchez M, Tischer T, Filardo G, Sabatier F, Magalon J. The Top 100 Most Cited Articles on Platelet-Rich Plasma Use in Regenerative Medicine-A Bibliometric Analysis-From the ESSKA Orthobiologic Initiative. Bioengineering (Basel). 2022 Oct 19;9(10):580. doi: 10.3390/bioengineering9100580. PMID 36290547
- [Background] Zheng Z, Yin J, Cheng B, Huang W. Materials Selection for the Injection into Vaginal Wall for Treatment of Vaginal Atrophy. Aesthetic Plast Surg. 2021 Jun;45(3):1231-1241. doi: 10.1007/s00266-020-02054-w. Epub 2021 Mar 1. PMID 33649927
- [Background] Ribeiro APL, Oliveira BGRB. Production cost of autologous platelet rich plasma gel. Rev Lat Am Enfermagem. 2019 Dec 5;27:e3221. doi: 10.1590/1518-8345.3265.3221. eCollection 2019. PMID 31826162
- [Background] Dougherty EJ. An evidence-based model comparing the cost-effectiveness of platelet-rich plasma gel to alternative therapies for patients with nonhealing diabetic foot ulcers. Adv Skin Wound Care. 2008 Dec;21(12):568-75. doi: 10.1097/01.ASW.0000323589.27605.71. PMID 19065083
- [Background] Marx RE. Platelet-rich plasma: evidence to support its use. J Oral Maxillofac Surg. 2004 Apr;62(4):489-96. doi: 10.1016/j.joms.2003.12.003. No abstract available. PMID 15085519
- [Background] Cho MJ, Rohrich RJ. Level of Evidence on Platelet-rich Plasma in Plastic Surgery. Plast Reconstr Surg Glob Open. 2021 Apr 15;9(4):e3379. doi: 10.1097/GOX.0000000000003379. eCollection 2021 Apr. PMID 33868870
- [Background] Sclafani AP, McCormick SA. Induction of dermal collagenesis, angiogenesis, and adipogenesis in human skin by injection of platelet-rich fibrin matrix. Arch Facial Plast Surg. 2012 Mar-Apr;14(2):132-6. doi: 10.1001/archfacial.2011.784. Epub 2011 Oct 17. PMID 22006233
- [Background] Alves R, Grimalt R. A Review of Platelet-Rich Plasma: History, Biology, Mechanism of Action, and Classification. Skin Appendage Disord. 2018 Jan;4(1):18-24. doi: 10.1159/000477353. Epub 2017 Jul 6. PMID 29457008
- [Background] Mantovani M, Gennai A, Russo PR. A new approach to regenerative medicine in gynecology. Int J Gynaecol Obstet. 2022 Jun;157(3):536-543. doi: 10.1002/ijgo.13906. Epub 2021 Sep 24. PMID 34463351
- [Background] Aguilar P, Hersant B, SidAhmed-Mezi M, Bosc R, Vidal L, Meningaud JP. Novel technique of vulvo-vaginal rejuvenation by lipofilling and injection of combined platelet-rich-plasma and hyaluronic acid: a case-report. Springerplus. 2016 Jul 26;5(1):1184. doi: 10.1186/s40064-016-2840-y. eCollection 2016. PMID 27512643
- [Background] Kim SH, Park ES, Kim TH. Rejuvenation Using Platelet-rich Plasma and Lipofilling for Vaginal Atrophy and Lichen Sclerosus. J Menopausal Med. 2017 Apr;23(1):63-68. doi: 10.6118/jmm.2017.23.1.63. Epub 2017 Apr 28. PMID 28523261
- [Background] Biglia N, Del Pup L, Masetti R, Villa P, Nappi RE. Vulvovaginal atrophy (VVA) in breast cancer survivors (BCS) is still an unmet medical need: results of an Italian Delphi Panel. Support Care Cancer. 2020 Jun;28(6):2507-2512. doi: 10.1007/s00520-019-05272-4. Epub 2020 Jan 22. PMID 31970513
- [Background] Nappi RE, Martini E, Cucinella L, Martella S, Tiranini L, Inzoli A, Brambilla E, Bosoni D, Cassani C, Gardella B. Addressing Vulvovaginal Atrophy (VVA)/Genitourinary Syndrome of Menopause (GSM) for Healthy Aging in Women. Front Endocrinol (Lausanne). 2019 Aug 21;10:561. doi: 10.3389/fendo.2019.00561. eCollection 2019. PMID 31496993
- [Background] Oyarzun MFG, Castelo-Branco C. Local hormone therapy for genitourinary syndrome of menopause in breast cancer patients: is it safe? Gynecol Endocrinol. 2017 Jun;33(6):418-420. doi: 10.1080/09513590.2017.1290076. Epub 2017 Feb 21. PMID 28277141
- [Background] Palma F, Volpe A, Villa P, Cagnacci A; Writing group of AGATA study. Vaginal atrophy of women in postmenopause. Results from a multicentric observational study: The AGATA study. Maturitas. 2016 Jan;83:40-4. doi: 10.1016/j.maturitas.2015.09.001. Epub 2015 Sep 14. PMID 26421474
- [Background] DiBonaventura M, Luo X, Moffatt M, Bushmakin AG, Kumar M, Bobula J. The Association Between Vulvovaginal Atrophy Symptoms and Quality of Life Among Postmenopausal Women in the United States and Western Europe. J Womens Health (Larchmt). 2015 Sep;24(9):713-22. doi: 10.1089/jwh.2014.5177. Epub 2015 Jul 22. PMID 26199981
- [Background] Tinelli A, Malvasi A, Rahimi S, Negro R, Vergara D, Martignago R, Pellegrino M, Cavallotti C. Age-related pelvic floor modifications and prolapse risk factors in postmenopausal women. Menopause. 2010 Jan-Feb;17(1):204-12. doi: 10.1097/gme.0b013e3181b0c2ae. PMID 19629013
- [Background] Ohta H, Hatta M, Ota K, Yoshikata R, Salvatore S. Online survey of genital and urinary symptoms among Japanese women aged between 40 and 90 years. Climacteric. 2020 Dec;23(6):603-607. doi: 10.1080/13697137.2020.1768236. Epub 2020 Jul 28. PMID 32720549
- [Background] Particco M, Djumaeva S, Nappi RE, Panay N, Palacios S; EVES Study investigators. The European Vulvovaginal Epidemiological Survey (EVES): impact on sexual function of vulvovaginal atrophy of menopause. Menopause. 2020 Apr;27(4):423-429. doi: 10.1097/GME.0000000000001496. PMID 32068686
- [Background] Nappi RE, de Melo NR, Martino M, Celis-Gonzalez C, Villaseca P, Rohrich S, Palacios S. Vaginal Health: Insights, Views & Attitudes (VIVA-LATAM): results from a survey in Latin America. Climacteric. 2018 Aug;21(4):397-403. doi: 10.1080/13697137.2018.1461826. Epub 2018 May 9. PMID 29741110
- [Background] Nappi RE, Palacios S, Panay N, Particco M, Krychman ML. Vulvar and vaginal atrophy in four European countries: evidence from the European REVIVE Survey. Climacteric. 2016 Apr;19(2):188-97. doi: 10.3109/13697137.2015.1107039. Epub 2015 Nov 19. PMID 26581580
- [Background] Szymanski J, Zareba K, Jakiel G, Slabuszewska-Jozwiak A. Genitourinary syndrome of menopause - is the problem solved? State of the art 2018. Prz Menopauzalny. 2018 Dec;17(4):168-174. doi: 10.5114/pm.2018.81741. Epub 2018 Dec 31. PMID 30766464
- [Background] Sturdee DW, Panay N; International Menopause Society Writing Group. Recommendations for the management of postmenopausal vaginal atrophy. Climacteric. 2010 Dec;13(6):509-22. doi: 10.3109/13697137.2010.522875. Epub 2010 Sep 30. PMID 20883118